CLINICAL TRIAL: NCT07381309
Title: Oncolytic Virus (H101) Peritumoral Injection Combined With SBRT, Chemotherapy, Targeted Therapy, and Immunotherapy for Unresectable MSS/pMMR Colorectal Cancer Liver Metastases (CRLM)
Brief Title: Oncolytic Virus (H101) + SBRT + Chemotherapy + Targeted Therapy + Immunotherapy for Unresectable CRLM
Acronym: VVSHIP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jun Huang (Other)
Responsible Party: Sponsor-Investigator, Jun Huang, Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Organization: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2025404
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: CRC; Liver Metastasis Colon Cancer
Keywords: Stereotactic body radiation therapy; Targeting Therapy; PD-1 Monoclonal Antibody; Oncolytic Virus
MeSH Terms: interventions — Radiosurgery; spartalizumab; Oncolytic Virotherapy; IFL protocol; Irinotecan; Leucovorin; Fluorouracil; Drug Therapy

STUDY DESIGN:
Masking Description: No mask
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- H101 + SBRT + PD-1 Antibody + Targeted Therapy + Chemotherapy (Experimental): The treatment regimen is administered sequentially as follows. Following stereotactic body radiotherapy (SBRT), a peritumoral injection of H101 is administered one week later. Three days after the H101 injection, combination therapy with chemotherapy and the PD-1 monoclonal antibody is initiated. This is followed by four cycles of a combined regimen consisting of peritumoral H101 injection, PD-1 monoclonal antibody, chemotherapy, and targeted therapy, with each cycle administered every 21 days.
  Interventions: Radiation: SBRT; Drug: PD-1 Antibody; Drug: H101; Drug: Target Therapy; Combination Product: Chemotherapy
- Folfiri + Targeted Therapy (Active Comparator): Patients will receive four cycles of the FOLFIRI chemotherapy regimen combined with targeted therapy selected based on genetic testing results, with each cycle administered every 21 days.
  Interventions: Drug: Target Therapy; Combination Product: FOLFIRI

INTERVENTIONS:
Radiation: SBRT — Stereotactic Body Radiotherapy
  Other Names: stereotactic body radiotherapy
  Arms: H101 + SBRT + PD-1 Antibody + Targeted Therapy + Chemotherapy
Drug: PD-1 Antibody — PD-1 Antibody every 21 days
  Other Names: PD-1 Monoclonic Antibody
  Arms: H101 + SBRT + PD-1 Antibody + Targeted Therapy + Chemotherapy
Drug: H101 — Peritumoral Injection of oncolytic virus (H101)
  Other Names: oncolytic virus
  Arms: H101 + SBRT + PD-1 Antibody + Targeted Therapy + Chemotherapy
Drug: Target Therapy — Targeted agents selected based on genetic testing results
  Other Names: Target agents
Combination Product: FOLFIRI — FOLFIRI is a standard biweekly chemotherapy regimen for metastatic colorectal cancer. It consists of irinotecan, leucovorin, and fluorouracil (5-FU) administered sequentially over a 46-hour infusion period per cycle.
  Other Names: irinotecan, leucovorin, and fluorouracil
  Arms: Folfiri + Targeted Therapy
Combination Product: Chemotherapy — Fluorouracil-based chemotherapy regimens, such as FOLFOX, CAPOX, or FOLFIRI.
  Other Names: Fluorouracil-based chemotherapy
  Arms: H101 + SBRT + PD-1 Antibody + Targeted Therapy + Chemotherapy

SUMMARY:
This prospective study aims to investigate the efficacy and safety of peritumoral injection of the oncolytic virus H101 in combination with stereotactic body radiotherapy (SBRT), PD-1 monoclonal antibody, chemotherapy, and targeted therapy for the treatment of patients with unresectable, microsatellite stable/mismatch repair proficient (MSS/pMMR) colorectal adenocarcinoma liver metastases. The ultimate goal is to provide high-level evidence-based medical support for this combined modality approach.

DETAILED DESCRIPTION:
Given the complexity and heterogeneity of the tumor microenvironment, the overall efficacy of monotherapy is limited, making combination therapy the prevailing trend in oncology. In recent years, comprehensive cancer treatment strategies have flourished, with targeted therapy, immunotherapy, and gene therapy being key research focuses. Oncolytic adenovirus stands out as one of the most promising directions in gene therapy. Clinical studies have found a synergistic effect between oncolytic adenovirus and PD-1 antibodies, establishing durable anti-tumor immunity. This suggests that the triple combination of an oncolytic virus (OV, e.g., H101), stereotactic body radiotherapy (SBRT), and a PD-1 monoclonal antibody may yield clinical benefits surpassing existing therapies. However, to date, there have been no clinical reports on the combination of H101, SBRT, and a PD-1 inhibitor for treating unresectable liver metastases.

Our institution previously conducted an exploratory treatment on a patient with unresectable colorectal cancer (CRC) liver metastases using a comprehensive regimen of SBRT (40 Gy in 5 fractions, BED=72 Gy) combined with peritumoral H101 injection and a PD-1 inhibitor. Follow-up exceeding one year showed a partial response (PR) on imaging evaluation, with no local progression in the liver metastases and the absence of grade ≥3 radiotherapy-related adverse events. This preliminary result demonstrates the potential efficacy and safety of this combination. Nevertheless, high-quality clinical evidence is still lacking to confirm whether patients with unresectable CRC liver metastases can derive further benefit from the H101+SBRT+PD-1 inhibitor regimen-such as improved objective response rate (ORR) and survival, or even achieving a no evidence of disease (NED) status in liver metastases for some patients-necessitating validation through prospective studies.

Based on the aforementioned background and preliminary exploration, we plan to conduct a multicenter, prospective, single-arm, phase II clinical study. It aims to evaluate the efficacy and safety of the H101 + SBRT + PD-1 inhibitor combination in patients with unresectable CRC liver metastases. This study will investigate whether this triple therapy can improve the ORR, reduce the local recurrence rate, potentially enable some patients to reach NED status, and consequently prolong disease-free survival (DFS). The study plans to enroll 114 participants over a trial period of 3 years, with the goal of providing high-level evidence-based medical support for this innovative combined regimen in treating unresectable CRC liver metastases.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or their legal representative understands and signs the informed consent form.
2. Patients with pMMR/MSS colorectal adenocarcinoma.
3. Aged 18-75 years.
4. Patients with histologically or cytologically confirmed colorectal cancer liver metastases. There must be at least one injectable lesion in the liver, which must also meet the criteria for a measurable target lesion according to RECIST version 1.1 (≥10 mm in the longest diameter on spiral CT/MRI scan with a slice thickness of no greater than 5 mm).
5. Patients with definitively unresectable metachronous liver metastases; OR patients deemed surgically resectable but who refuse surgery, provided the liver metastases meet the following requirements: ① The number of metastatic lesions must be no more than 5, and the sum of the longest diameters of all metastatic lesions must be ≤100 mm; ② The longest diameter of a single lesion must be ≤100 mm; ③ The longest diameter of the lesion to be injected must be ≥10 mm and ≤80 mm.
6. The liver metastases have not received prior radiotherapy, OR the area of the liver near the planned radiotherapy site has not been previously irradiated. At least 700 cc of liver volume must be preserved outside the treatment area.
7. Prior treatments such as hepatic resection, systemic chemotherapy, local ablation therapy, or hepatic artery infusion pump chemotherapy are allowed, provided a washout period of 2 weeks is observed. Patients must have recovered from prior anti-tumor therapy-related adverse events to baseline or Grade ≤1 (according to CTCAE version 5.0) (excluding alopecia and Grade 2 anemia).
8. Child-Pugh score A or B
9. ECOG Performance Status 0-1
10. Peripheral blood counts and liver/renal function within the allowable ranges (tested within 15 days before treatment initiation)
11. No prior history of other concomitant malignancies. Patients must not be pregnant or breastfeeding and should use effective contraception during the study and for 6 months after the last dose.
12. Life expectancy ≥6 months.

Exclusion Criteria:

1. Synchronous colorectal cancer liver metastases.
2. Active hepatitis, cirrhosis, or Child-Pugh class C.
3. Extralepatic metastases to: central nervous system / bone marrow / brain (UICC 8th edition).
4. Liver metastases not measurable.
5. Prior history of oncolytic virus therapy (e.g., T-VEC).
6. Liver metastases not meeting the requirements for peritumoral injection volume or unsuitable for peritumoral injection.
7. History of severe drug allergy (e.g., to oncolytic adenovirus, PD-1 monoclonal antibody, platinum agents, 5-FU, leucovorin, 5-HT3 receptor antagonists, bevacizumab, etc.).
8. Antiviral therapy (e.g., acyclovir, ganciclovir, valacyclovir, vidarabine) within 4 weeks prior to the first dose of study treatment.
9. Participation in another clinical trial within 4 weeks or ongoing participation.
10. History of prior therapy targeting PD-1, PD-L1, PD-L2, CTLA-4, or any other T-cell co-stimulation or checkpoint pathway.
11. Severe electrolyte abnormalities.
12. Significant portal hypertension: history of upper gastrointestinal bleeding or severe hypersplenism.
13. Arterial or deep venous thrombosis within the past 6 months; history or evidence of bleeding tendency within the past 2 months.
14. Pregnant or breastfeeding women, or women with a positive pregnancy test before the first dose; or female participants and their partners unwilling to use strict contraception during the study.
15. Active autoimmune disease requiring systemic treatment (e.g., immunomodulators, corticosteroids, immunosuppressants) within the past 2 years.
16. Past or current other active malignancies (except malignancies cured >3 years ago or carcinoma in situ treated curatively).
17. Severe ECG abnormalities; active coronary artery disease, severe/unstable angina, newly diagnosed angina, or myocardial infarction within 12 months; New York Heart Association (NYHA) class II or higher congestive heart failure.
18. Active infection (with fever >38°C).
19. Poorly controlled hypercalcemia, hypertension, or diabetes.
20. Severe pulmonary disease (interstitial pneumonia, pulmonary fibrosis, severe emphysema, etc.).
21. Psychiatric disorder affecting clinical treatment or history of central nervous system disease.
22. Severe complications (intestinal obstruction, renal insufficiency, hepatic insufficiency, cerebrovascular disorders, etc.).
23. Persistent toxicity ≥ Grade 2 (CTCAE v5.0) from prior therapy (except anemia, alopecia, skin pigmentation).
24. Use of any other investigational drug or participation in another interventional trial within 14 days prior to study treatment.
25. Pregnant, breastfeeding, or planning pregnancy during the study; men or women unwilling to use effective contraception.
26. Any unstable medical condition that may affect patient safety or compliance, as judged by the investigator to be unsuitable for the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 year
  Objective Response Rate

SECONDARY OUTCOMES:
1 year PFS | 1 year
  1 year Progression Free Survival
1 year OS | 1 year
  1 year Overall Survival
R0 Resection Rate | 1 year
  R0 Resection Rate
pCR | 1 year
  Pathological Complete Response
DCR | 1 year
  Disease Control Rate
AE rate | 1 year
  Adverse Event rate

CONTACTS AND LOCATIONS:
Overall Officials: Jun Huang, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No